CLINICAL TRIAL: NCT00122928
Title: Environmental Approaches for Obesity Management at Dow
Brief Title: Comparison of Workplace Obesity Management Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ron Goetzel, Research Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00009301; R01HL079546 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Obesity; Cardiovascular Diseases; Heart Diseases
Keywords: Worksite; Workplace; Return on Investment; Financial Impact
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Heart Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High intensity environmental intervention (Experimental): Intense intervention
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Environmental Obesity Program - Healthy Culture
- Moderate intensity environmental intervention (Experimental): Moderate intervention
  Interventions: Behavioral: Diet; Behavioral: Exercise
- Individual intervention only (No Intervention): Control

INTERVENTIONS:
Behavioral: Diet — Healthy Choices in vending machines; Healthy Choices in cafeteria; Catering (Healthy Choices in site meetings, shutdowns, OT meals, etc.); Targeted Messages: Nutrition; Site Based Rewards and Recognition - Individual Employees Weight Management Tracking Program
  Arms: High intensity environmental intervention; Moderate intensity environmental intervention
Behavioral: Exercise — Walking Paths/Routes; Weight Management Tracking Program; Targeted Messages: Physical Activity; Site Based Rewards and Recognition - Individual Employees
  Arms: High intensity environmental intervention; Moderate intensity environmental intervention
Behavioral: Environmental Obesity Program - Healthy Culture — Site Goal Setting; Work Group Alignment to Site Goals; Reporting to Senior Leadership; Leadership Training; Site Leadership, Cross Discipline Teams, Work Groups, Healthy Culture Focal Point Rewards and Recognition
  Arms: High intensity environmental intervention

SUMMARY:
The purpose of this study is to design and demonstrate the feasibility of implementing moderate and intensive environmental obesity prevention programs at major worksites.

DETAILED DESCRIPTION:
BACKGROUND:

More than half of all Americans are overweight or obese, and the prevalence of these risk factors has increased dramatically in the past decade. Obesity is a risk factor for several chronic illnesses, including type 2 diabetes and heart disease. The national medical cost that is attributed to obesity is estimated to be between $60 and $93 billion. Business leaders are becoming increasingly aware of the human and economic burden that poor health imposes on their workers. Many employers have invested in health promotion and disease prevention programs aimed at reducing the prevalence of obesity in the workplace through the encouragement of physical activity, maintaining a healthy diet, and improved management of health risk factors. Employers continue to seek innovative and evidence-based programs that can be implemented in the workplace to address a growing public health epidemic that also adversely affects worker productivity.

DESIGN NARRATIVE:

The primary objective of this study will be to evaluate the effect of introducing two levels of environmental programs, in addition to existing individualized programs, at reducing obesity in the workplace. Five outcomes will be evaluated: 1) body mass index and other weight-related biometric measures; 2) behavioral health risk factors; 3) weight-related health conditions; 4) health care utilization and medical expenditures; and 5) employee productivity measured in terms of reduced absenteeism and on-the-job presenteeism. The study will also include an assessment of costs and benefits of the two programs, including the medical, absenteeism, and productivity benefits, and an assessment of the impact of the programs on the worksite climate. Twelve Dow chemical companies will participate in the study. Participants will be randomly assigned to a moderate environmental program, an intensive environmental program, or a control group, which will receive individualized treatment only. The moderate program will include inexpensive environmental changes (e.g., prompts and reminders). In the high intensity program, senior managers will assist in the development of a worksite culture that is broadly supportive of improved weight and health management by employees. Annual health screening and biometrics data along with administrative medical claims, absence records, and productivity survey data will be analyzed to determine program impacts. Non-experimental statistical methods will be used to control the differences that remain across sites after randomization. The study will also produce extensive information about how employers can successfully implement environmental programs to reduce obesity at worksites.

ELIGIBILITY:
Inclusion Criteria:

* Active employees at any of 12 participating company locations of The Dow Chemical Company
* Participants must be must be between 18 and 70 years old

Exclusion Criteria:

* The Dow Chemical Company employees located at a facility other than one of the 12 study sites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5124 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of obesity | Measured at baseline and at the end of years 1 and 2
Weight-related risk factors | Measured at baseline and at the end of years 1 and 2
Overall health and well-being | Measured at baseline and at the end of years 1 and 2
Healthcare utilization and expenditures | Measured at baseline and at the end of years 1 and 2
Employee productivity measures (i.e., absenteeism and presenteeism) | Measured at baseline and at the end of years 1 and 2
Return on investment (measured at Year 2) | Measured at baseline and at the end of years 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Ron Z. Goetzel, PhD, Principal Investigator — Emory University

REFERENCES:
- [Background] Goetzel RZ, Ozminkowski RJ, Baase CM, Billotti GM. Estimating the return-on-investment from changes in employee health risks on the Dow Chemical Company's health care costs. J Occup Environ Med. 2005 Aug;47(8):759-68. doi: 10.1097/01.jom.0000172868.05935.67. PMID 16093925
- [Background] Pratt CA, Lemon SC, Fernandez ID, Goetzel R, Beresford SA, French SA, Stevens VJ, Vogt TM, Webber LS. Design characteristics of worksite environmental interventions for obesity prevention. Obesity (Silver Spring). 2007 Sep;15(9):2171-80. doi: 10.1038/oby.2007.258. PMID 17890484
- [Background] Wilson MG, Goetzel RZ, Ozminkowski RJ, DeJoy DM, Della L, Roemer EC, Schneider J, Tully KJ, White JM, Baase CM. Using formative research to develop environmental and ecological interventions to address overweight and obesity. Obesity (Silver Spring). 2007 Nov;15 Suppl 1(Suppl 1):37S-47S. doi: 10.1038/oby.2007.386. PMID 18073340
- [Background] Della LJ, DeJoy DM, Goetzel RZ, Ozminkowski RJ, Wilson MG. Assessing management support for worksite health promotion: psychometric analysis of the leading by example (LBE) instrument. Am J Health Promot. 2008 May-Jun;22(5):359-67. doi: 10.4278/ajhp.22.5.359. PMID 18517097
- [Background] Dejoy DM, Wilson MG, Goetzel RZ, Ozminkowski RJ, Wang S, Baker KM, Bowen HM, Tully KJ. Development of the Environmental Assessment Tool (EAT) to measure organizational physical and social support for worksite obesity prevention programs. J Occup Environ Med. 2008 Feb;50(2):126-37. doi: 10.1097/JOM.0b013e318161b42a. PMID 18301169
- [Background] Goetzel RZ, Bowen J, Ozminkowski RJ, Kassed, C, Roemer, EC, Tabrizi MJ, Short M, Wang S, Pei X, Bowen H, DeJoy DM, Wilson MG, Baker K, Tully K, White JM, Billotti GM, Baase CM (In press). Case Study: Introducing Environmental Interventions at The Dow Chemical Company Aimed at Reducing Overweight and Obesity among Workers. Book chapter in American College of Sports Medicine Worksite Health Handbook. Second Edition: Healthy Worker, Healthy Company, Pronk N (ed.) Human Kinetics.
- [Background] Goetzel RZ, Baker KM, Short ME, Pei X, Ozminkowski RJ, Wang S, Bowen JD, Roemer EC, Craun BA, Tully KJ, Baase CM, DeJoy DM, Wilson MG. First-year results of an obesity prevention program at The Dow Chemical Company. J Occup Environ Med. 2009 Feb;51(2):125-38. doi: 10.1097/JOM.0b013e3181954b03. PMID 19209033